CLINICAL TRIAL: NCT00380510
Title: The SAFE TEEN Study: Family Physicians' Reports of Facilitators of and Barriers to Preventive Care for Adolescents.
Brief Title: The Safe Teen Study
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Other Study IDs: HP000016-02
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2006-09-26 (Estimated); Status verified 2006-09

CONDITIONS: Prevention
Keywords: Family Physicians; Adolescents; Preventive Care; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The study examines (1)the incidence of preventive health services provided by family physicians to adolescent patients, and (2)barriers and facilitators of prevention discussions between family physicians and their adolescent patients.

DETAILED DESCRIPTION:
This study used a card study design to allow volunteer physicians to record research data in the context of providing clinical care. The method was brief, simple, and convenient for busy practicing clinicians.

Volunteer resident physicians and faculty carried data collection checklists in their pockets and completed one for every adolescent patient seen during a randomly selected two week period. Physicians attempted to collect data on ten consecutive encounters with teen patients aged 11-21 years. The checklist documented patient characteristics (age, gender and ethnicity), reason for visit, parent presence, and types of prevention issues discussed during the visit. Patient and visit information was collected to assess its influence on physician prevention discussions. Finally, the checklist asked open-ended questions related to barriers to and facilitators to teen prevention discussions.

The study involved five clinical sites comprising approximately 140 faculty and resident family physicians. The investigators sought 10-15 volunteer physicians from each site (60-90 physicians), and asked them to complete data checklists on 10 consecutive adolescent patients (600-900 visits). After a training session, each site randomly selected data collection periods.

Physicians provided usual care for adolescent patients and recorded on the checklists any prevention discussions during the visit.

ELIGIBILITY:
Inclusion Criteria:

* Family Medicine Residency physicians and faculty in six residency programs in Texas

Exclusion Criteria:

* Physicians not in the residency programs

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-06; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K Burge, Ph.D., Principal Investigator — University of TexasHealth Science Center at San Antonio
Locations (5):
- United States (5):
  - Christus Memorial Hospital Spohn Family Medicine Residency Program, Corpus Christi, Texas
  - Valley Baptist Family Medicine Program, Harlingen, Texas
  - McAllen Family Medicine Residency Program, McAllen, Texas
  - Family Medicine Residency Program, Christus Santa Rosa Hospital, San Antonio, Texas
  - Department of Family and Community Medicine UTHSCSA, San Antonio, Texas